CLINICAL TRIAL: NCT01438333
Title: Efficacy of INERSAN in Patients With Chronic Periodontitis as Adjunctive to Full Mouth Disinfection: a Randomized, Double Masked, Placebo Controlled Clinical Trial
Brief Title: Efficacy of INERSAN in Patients With Chronic Periodontitis as Adjunctive to Full Mouth Disinfection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, Adjunct Professor, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07/CE/2011
Record Dates: First submitted 2011-09-13; First posted 2011-09-22 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Peridodontitis; probiotics; lactobacillus brevis; full mouth disinfection
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus brevis (Experimental)
  Interventions: Dietary Supplement: lactobacillus brevis tablets
- Placebo (Placebo Comparator): 5 tablets a day for 6 weeks
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: lactobacillus brevis tablets — 5 tablets a day for 6 weeks
  Other Names: Inersan
  Arms: Lactobacillus brevis
Dietary Supplement: PLACEBO — 5 tablets a day for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate beneficial effects of probiotic Lactobacillus brevis CD2 tablets in addition to the primary treatment for patients with chronic periodontitis (Full Mouth Disinfection), at local level and at systemic level.

DETAILED DESCRIPTION:
This study will be conducted as a double blind, randomized, parallel group, placebo controlled clinical trial, involving subjects of 21 years of age or older to evaluate the beneficial effects of INERSAN® tablets as the primary treatment for patients with chronic periodontitis.

Patients satisfying the "Inclusion criteria" will be enrolled into the study after explaining them the objective of the study and after taking their written consent.

The probiotic tablets used in the present study contain a single strain of Lactobacilli, Lactobacillus brevis CD2, as active component. The placebo will be a mix of sugars and salts used as excipients in the active formulation. The active study medication and Placebo will be identical in appearance and organoleptic properties. Study treatment will be started from the day of enrollment and continued for 6 weeks. The daily dose of trial product will be 5 tablets per day, one tablet to be taken every 2-3 hours. The tablets will be to be kept in mouth for it to dissolve by itself. A hot beverage (e.g.: tea, coffee, milk etc.) will not to be taken for at least half an hour before and after the medication since elevated temperature could inactivate the bacteria.

The study drug and placebo will be provided as per the randomization schedule, packed in patient specific packs, bearing patient number. The study being a double masked study, both the patient and the Investigator will be blinded during the entire course of the trial. A sealed copy of the randomization codes will be given to the Principal Investigator and will be directed to open and break the codes only at the event of adverse events after discussion with sponsor and the monitor.

Patients will be informed that they may withdraw from the study at any time for any reasons. The Investigator also has the right to withdraw patients from the study if it is in the best interest of the patient. The reason and date of discontinuation will to be clearly documented in the case report form for all patients who discontinued the study product prematurely.

Periodontal examination periodontal probe depth (PPD), clinical attachment level (CAL), bleeding on probing index (BOP),plaque index (PI), and tooth mobility, will be conducted at the screening period and scheduled study visits. Photographs of the dental cavity were taken at the start and end of the study treatment.

Radiographs were compared at the beginning and end of the study to compare the bone level and record other relevant findings.

At baseline each volunteer will be received a Full Mouth Disinfection (FMD) and, to ensure that all deposits has been removed, a disclosing episode will be carried out after which any remaining plaque will be removed.

Saliva samples (at least 3 mL) will be collected in eppendorf tubes and immediately frozen at -20°C.

The activity of Arginine deiminase will be evaluated by High Performance Liquid Chromatography of fluorescence derivatized aminoacids, by monitoring the formation of citrulline from Arginine.

For metabonomic analysis the saliva samples will be collected in the morning in a sterile tube containing sodium fluoride as an antimicrobic agent. Patients must refrain from eating, drinking, smoking or dental washing before the collection.

The samples will be kept on ice and will be stored at -80°C as soon as possible.

Plaque samples will be collected with a sterile curette and dispersed in sterilized saline solution and stored at -20°C.

Microbiota will be analyzed on DNA extracted from the samples using a Qiagen kit. L.brevis CD2 strain will be detected using a TaqMan Real Time PCR, by using specifically designed primers. Microbial flora potentially involved in periodontitis, will be identified and quantified by molecular biology techniques.

Breath samples will be collected in 1 mL disposable syringe (latex-free) and immediately analyzed between a portable gas chromatograph device (Oral Chroma, Abimedical corporation, Osaka, Japan).

Blood samples (20-25mL) will be collected by only 20% of population on the study al baseline and at end of the treatment period (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 21-70 years of age groups;
* patients with chronic periodontitis in need of primary treatment;
* patients with at least 20 fully erupted teeth;
* patients ready to give written informed consent for participating in the trial;
* patients agreeing to comply with the study protocol and instructions.

Exclusion Criteria:

* Pregnant women and lactating mothers;
* patients with debilitating systemic diseases;
* patients in needs for prophylactic antibiotics;
* patients treated with antibiotics within 30 days prior to enrollment into the study;
* patients already participant any other clinical trial or participant other investigational drug, or food supplement, in the last 30 days;
* patient having active periapical abscess or periodontal abscess or a history of acute necrotizing ulcerative gingivitis;
* patients not willing to participate in the trial.
* patients with psychiatric problems.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparison in saliva and gingival crevicular fluid samples of the levels of Matrixmetalloproteinases (MMPs) | 6 weeks
Comparison in saliva and gingival crevicular fluid samples of the levels of modulators of inflammatory reaction (interleukin 1beta, interleukin 10, prostaglandin 2) | 6 weeks
Comparison in saliva samples of the levels of metabolic phenotype | 6 weeks

SECONDARY OUTCOMES:
Comparison in saliva samples of the levels of Nitric Oxide Synthase (NOS) activity; | 6 weeks
Comparison in saliva samples of the levels of Arginine deiminase | 6 weeks
Comparison in saliva samples of the levels of lactoferrin | 6 weeks
Comparison in saliva and gingival crevicular fluid samples of the levels of subgingival bacteria (Aggregatibacter Actinomycetemcomitan, Porphyromonas gingivalis, Tannerella Forsythia, Treponema denticola) | 6 weeks
Comparison in breath samples of the levels of Volatile Sulfur Compounds (VSC)(hydrogen sulfide, methyl mercaptan, dimethyl sulfide) | 6 weeks
Comparison in blood samples of the levels of Toll Like Receptor-2 and Toll Like Receptor-4 positive B-cells | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ENRICO MARCHETTI, DDS, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, Division of Periodontology, L’Aquila, AQ, Italy